CLINICAL TRIAL: NCT00675012
Title: NGR005: Pilot Study of NGR-hTNF Administered at Low and High Doses in Combination With a Standard Oxaliplatin Based Regimen in Patients With Metastatic Colorectal Cancer
Brief Title: NGR-hTNF Administered in Combination With a Standard Oxaliplatin Based Regimen in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR005; 2007-003668-24 (EudraCT Number)
Record Dates: First submitted 2008-05-05; First posted 2008-05-08 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Colon Cancer
Keywords: NGR-hTNF; Capecitabine; Oxaliplatin; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: NGR-hTNF; Drug: Oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: NGR-hTNF — iv 0.8 or 45 mcg/sqm q3W
Drug: Oxaliplatin — iv q3W 100 mg/sqm 60 minutes after NGR-hTNF infusion
Drug: capecitabine — orally 825 mg/sqm 2qDx14

SUMMARY:
The main objective of the trial is to document the safety of NGR-hTNF administered at low and high doses in combination with a standard oxaliplatin based regimen in patients with metastatic colorectal cancer not amenable to any clinical improvement by current standard treatments

DETAILED DESCRIPTION:
Phase II, open-label, non-randomized study that will be conducted in two sequential cohorts of patients. Patients with metastatic colorectal cancer not amenable to any clinical improvement by current standard treatments are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with metastatic colorectal cancer (CRC) treated with no more than three standard systemic regimens (including biologic agents) for metastatic disease
* Life expectancy more than 3 months
* ECOG Performance status 0-1
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils >1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin <1.5 x ULN
  * AST and/or ALT <2.5 x ULN in absence of liver metastasis
  * AST and/or ALT <5 x ULN in presence of liver metastasis
  * Serum creatinine <1.5 x ULN
  * Creatinine clearance (estimated according to Cockcroft-Gault formula) ≥ 50 ml/min
* Patients may have had prior therapy providing the following conditions are met:

  * Chemotherapy, radiation therapy, hormonal therapy or immunotherapy: wash-out period of 28 days before start treatment
  * Surgery: wash-out period of 14 days before start treatment
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients must not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Uncontrolled hypertension
* Prolonged QTc interval (congenital or acquired)
* Patient with significant peripheral vascular disease
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Symptomatic peripheral neuropathy ≥ grade 1 according the NCI CTCAE v.3.0.
* Known hypersensitivity/allergic reaction or contraindications to human albumin preparations or to any of the excipients
* Known hypersensitivity/allergic reaction or contraindications to platinum compounds or fluoropyrimidines
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation.
* Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study.
* Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and safety of NGRhTNF administered at low (0.8 mcg/sqm) and high (45 mcg/sqm) doses in combination with a standard oxaliplatin-based regimen in two sequential cohorts of patients with metastatic colorectal cancer. | during the study

SECONDARY OUTCOMES:
Document the preliminary antitumor activity in terms of objective response rate (according to RECIST criteria) and progression-free survival | during the study
Evaluate the pharmacokinetic profile of NGRhTNF and to measure plasma levels of sTNF-RI and sTNF-RII | before during and following the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sobrero, MD, Principal Investigator — Azienda Ospedaliera Universitaria San Martino Genoa, Italy
Locations (1):
- Azienda Ospedaliera Universitaria San Martino, Genoa, Genoa, Italy

REFERENCES:
- [Result] Mammoliti S, Andretta V, Bennicelli E, Caprioni F, Comandini D, Fornarini G, Guglielmi A, Pessino A, Sciallero S, Sobrero AF, Mazzola G, Lambiase A, Bordignon C. Two doses of NGR-hTNF in combination with capecitabine plus oxaliplatin in colorectal cancer patients failing standard therapies. Ann Oncol. 2011 Apr;22(4):973-978. doi: 10.1093/annonc/mdq436. Epub 2010 Sep 20. PMID 20855468